CLINICAL TRIAL: NCT02610881
Title: Acceptability and Feasibility of Micronutrient Powders Versus Iron Syrup for Anemia Prevention in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: International Food Policy Research Institute (Other)
Responsible Party: Principal Investigator, Melissa Fox Young, Research Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: IRB00081930
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Iron; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iron and Folic Acid (IFA)/Micronutrient Powders (MNP) (Experimental): Participants will receive iron and folic acid (IFA) drops for one month followed by a two week washout period. Participants will then receive micronutrient powders (MNP) for one month. Mothers of participants will receive counseling on the benefits of iron intake, side effects of IFA, and preservation of IFA bottles and MNP sachets.
  Interventions: Dietary Supplement: Iron and Folic Acid (IFA); Dietary Supplement: Micronutrient Powders (MNP); Behavioral: Iron Plus Strategy Counseling
- Micronutrient Powders (MNP)/Iron and Folic Acid (IFA) (Experimental): Participants will receive micronutrient powders (MNP) for one month followed by a two week washout period. Participants will then receive iron and folic acid (IFA) drops for one month. Mothers of participants will receive counseling on the benefits of iron intake, side effects of IFA, and preservation of IFA bottles and MNP sachets.
  Interventions: Dietary Supplement: Iron and Folic Acid (IFA); Dietary Supplement: Micronutrient Powders (MNP); Behavioral: Iron Plus Strategy Counseling

INTERVENTIONS:
Dietary Supplement: Iron and Folic Acid (IFA) — 1 mg of IFA syrup (containing 20 mg of elemental iron and 100 mcg of folic acid) will be taken twice per week for one month.
Dietary Supplement: Micronutrient Powders (MNP) — One sachet of micronutrient powder will be mixed into food to be taken once daily for a total of one month. One sachet of micronutrient powders includes the following:
  Iron (Ferrous Fumarate) 12.5 mg Zinc (Zinc Gluconate) 5 mg Folic Acid 0.160 mg Vitamin-A (Vit-A Acetate) 0.30mg Vitamin-C (Ascorbic Acid) 30 mg Vitamin-B12 0.9 mcg Iodine 90 mcg Maltodextrin Base
Behavioral: Iron Plus Strategy Counseling — Mothers of participants will receive counseling on the benefits of regular iron intake, side effects associated with IFA administration, and the preservation of the IFA bottle and MNP sachets.

SUMMARY:
This study seeks to assess the acceptability, compliance, and preference for iron supplementation; micronutrient powders (MNP) versus iron syrup. Additionally, this study seeks to assess front line health worker perceptions and experiences regarding ease of implementation of each strategy and delivery strategy preference.

DETAILED DESCRIPTION:
The specific aims of this study are to assess the acceptability of, compliance, and preference for two delivery vehicles for pediatric prophylaxis iron supplementation (micronutrient powders (MNP) that contain iron versus iron syrup) among rural households in Bihar India delivered through home visits by front line health workers. Additionally, this study seeks to assess front line health worker perceptions and experiences regarding ease of implementation of each strategy and delivery strategy preference.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Children or one child per home

Exclusion Criteria:

* Currently taking iron supplements
* Mid upper arm circumference (MUAC) or less than 11.5 cm
* Suspected severe anemia
* Known case of haemoglobinopathy
* History of repeated blood transfusion
* Current pneumonia
* Current fever
* Acute diarrhea

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2015-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Acceptability of iron and folic acid (IFA) syrup | Endline (Up to 5 months)
  Caregiver change in acceptability of iron and folic acid (IFA) syrup will be assessed using the Relative Preference, Acceptability, and Compliance of Iron Syrup versus Multiple Micronutrient Powders (MMP) Among Infants 6-23 Months in Bihar, India survey. This survey collects information regarding the use of iron and nutrient supplementation, barriers to usage, and attitudes towards usage.
Acceptability of micronutrient powders (MNP) | Endline (Up to 5 months)
  Caregiver change in acceptability of micronutrient powders (MNP) will be assessed using the Relative Preference, Acceptability, and Compliance of Iron Syrup versus Multiple Micronutrient Powders (MMP) Among Infants 6-23 Months in Bihar, India survey. This survey collects information regarding the use of iron and nutrient supplementation, barriers to usage, and attitudes towards usage.
Preference for vitamin supplementation | Endline (Up to 5 months)
  Caregiver change in preference for vitamin supplementation (IFA versus MNP) will be assessed using the Relative Preference, Acceptability, and Compliance of Iron Syrup versus Multiple Micronutrient Powders (MMP) Among Infants 6-23 Months in Bihar, India survey. This survey collects information regarding the use of iron and nutrient supplementation, barriers to usage, and attitu
Vitamin supplementation compliance | Baseline, Endline (Up to 5 months)
  Caregiver change in vitamin supplementation compliance will be assessed using the Relative Preference, Acceptability, and Compliance of Iron Syrup versus Multiple Micronutrient Powders (MMP) Among Infants 6-23 Months in Bihar, India survey. This survey collects information regarding the use of iron and nutrient supplementation, barriers to usage, and attitudes towards usage.

SECONDARY OUTCOMES:
Change in perceived barriers to vitamin supplementation | Baseline, Endline (Up to 5 months)
  Caregiver change in perceived barriers to vitamin supplementation will be assessed using the Relative Preference, Acceptability, and Compliance of Iron Syrup versus Multiple Micronutrient Powders (MMP) Among Infants 6-23 Months in Bihar, India survey. This survey collects information regarding the use of iron and nutrient supplementation, barriers to usage, and attitudes towards usage.
Preferred method of distribution | Endline (Up to 5 months)
  The preferred method of distribution will be discussed with front line workers in focus group discussions.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Young, PhD, Principal Investigator — Emory University
Locations (1):
- CARE-India, Patna, Bihar, India

REFERENCES:
- [Derived] Young MF, Girard AW, Mehta R, Srikantiah S, Gosdin L, Menon P, Ramakrishnan U, Martorell R, Avula R. Acceptability of multiple micronutrient powders and iron syrup in Bihar, India. Matern Child Nutr. 2018 Apr;14(2):e12572. doi: 10.1111/mcn.12572. Epub 2017 Dec 6. PMID 29210507